CLINICAL TRIAL: NCT03406975
Title: Multi-center ESG Randomized Interventional Trial (MERIT-Trial)
Brief Title: Multicenter Endoscopic Sleeve Gastrectomy (ESG) Trial (MERIT Trial)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: University of Texas (Other); Johns Hopkins University (Other); Brigham and Women's Hospital (Other); Endeavor Health (Other); University of Chicago (Other); Orlando Health, Inc. (Other); Cornell University (Other); Avera McKennan Hospital & University Health Center (Other)
Responsible Party: Principal Investigator, Barham K. Abu Dayyeh, M.D., Barham Abu Dayyeh, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 17-007934
Record Dates: First submitted 2018-01-16; First posted 2018-01-23 (Actual); Results first posted 2022-10-18 (Actual); Last update posted 2022-10-18 (Actual); Status verified 2022-09

CONDITIONS: Obesity; Hypertension; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Obesity; Hypertension; Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (3):
- Control Group: Lifestyle Modification (Active Comparator): Participants randomized to the control group (lifestyle modification only) in Year 1 will undergo a standard moderate intensity life-style intervention during the first 12 months of participation.
  Interventions: Behavioral: Lifestyle Intervention
- Treatment Group: Overstitch ESG Procedure (Experimental): Participants randomized to the treatment group will proceed to have the Overstitch Endoscopic Sleeve Gastroplasty (ESG) at the start of Year 1 and will undergo a standard moderate intensity life-style intervention during the first 12 months of participation. All patients undergoing ESG will go on a 6 weeks transitional diet.ESG patients will undergo a standard moderate intensity life-style intervention administered over 15 12 visits in the first year after ESG. ESG patients who have not achieved >25% EWL at the end of Year 1 will undergo a repeat upper endoscopy at 52 to 60 weeks to assess the durability of the plications. Patients will continue follow-up with a modified lifestyle intervention program administered over 6 visits in the second year
  Interventions: Device: Overstitch Endoscopic Suture System; Behavioral: Lifestyle Intervention
- Crossover Group: Lifestyle Intervention to ESG Procedure (Experimental): Control group participants (lifestyle modification only) who were compliant with at least 75% of visits in Year 1, have not achieved ≥25% EWL or have a BMI >30 measured at the week 52 visit, and have no new psychosocial contraindications as deemed by the treatment team to the procedure will cross over to receive the Overstitch ESG in Year 2, in addition to the standard moderate intensity lifestyle intervention program of 12 months.
  Interventions: Device: Overstitch Endoscopic Suture System; Behavioral: Lifestyle Intervention

INTERVENTIONS:
Device: Overstitch Endoscopic Suture System — Endoscopic Sleeve Gastroplasty (ESG), an endoscopic minimally-invasive weight loss procedure, utilizing a suturing device to reduce the stomach volume by 80% through the creation of sleeve. This is accomplished by a series of endoscopically placed stitches through the stomach wall.
  Arms: Crossover Group: Lifestyle Intervention to ESG Procedure; Treatment Group: Overstitch ESG Procedure
Behavioral: Lifestyle Intervention — Standard low-calorie diet plan and moderate intensity life-style intervention of 150 minutes of aerobic exercise per week for 12 months.

SUMMARY:
Endoscopic Sleeve Gastroplasty (ESG) is an endoscopic minimally invasive weight loss procedure where a commercially available, FDA approved, full-thickness endoscopic suturing device (Overstitch; Apollo Endosurgery, Austin, TX) is used to reduce the stomach volume by 80% through the creation of a restrictive endoscopic sleeve. This is accomplished by a series of endoscopically placed full-thickness sutures through the gastric wall, extending from the antrum to the gastroesophageal junction.

Up to 200 participants at 9 locations in the United States will participate in this study.

The ESG procedure has been performed clinically since 2013 in the United States. The investigators are completing this study to compare how effective the ESG is for achieving long-term weight loss when compared to lifestyle modification only, as well as to evaluate the long-term safety and durability of the procedure and its impact on quality of life. Results of this research may help support having this procedure covered by health insurance plans for future patients.

ELIGIBILITY:
INCLUSION CRITERIA

1. Age 21-65
2. BMI ≥ 30 and ≤40 kg/m²
3. Willingness to comply with the substantial lifelong dietary restrictions required by the procedure
4. History of failure with non-surgical weight-loss methods
5. Willingness to follow protocol requirements, including signed informed consent, routine follow-up schedule, completing laboratory tests, and completing diet counseling
6. Residing within a reasonable distance from the investigator's office and able to travel to the investigator to complete all routine follow- up visits
7. Ability to give informed consent
8. Women of childbearing potential (i.e., not post-menopausal or surgically sterilized) must agree to use adequate birth control methods
9. ***There will be a quota for at least a) 50 patients with hypertension on one or more anti-hypertensive medication, b) 50 patients with type II diabetes mellitus on oral agents only with HgA1c ≤ 9, and thus the cohort of 200 patients will be stratified into three groups (Obesity, Obesity HTH, Obesity DM) and block randomized. No more than 50 participants without comorbidities will be enrolled in the trial.

EXCLUSION CRITERIA

1. History of foregut or gastrointestinal (GI) surgery (except uncomplicated cholecystectomy or appendectomy)
2. Prior gastrointestinal surgery with sequelae, i.e. obstruction, and/or adhesive peritonitis or known abdominal adhesions.
3. Prior open or laparoscopic bariatric surgery.
4. Prior surgery of any kind on the esophagus, stomach or any type of hiatal hernia surgery.
5. Any inflammatory disease of the gastrointestinal tract including esophagitis, Barrett's esophagus, gastric ulceration, duodenal ulceration, cancer or specific inflammation such as Crohn's disease.
6. Potential upper gastrointestinal bleeding conditions such as esophageal or gastric varices, congenital or acquired intestinal telangiectasis, or other congenital anomalies of the gastrointestinal tract such as atresias or stenoses.
7. A gastric mass or gastric polyps > 1 cm in size.
8. A hiatal hernia > 4cm of axial displacement of the z-line above the diaphragm or severe or intractable gastro-esophageal reflux symptoms.
9. A structural abnormality in the esophagus or pharynx such as a stricture or diverticulum that could impede passage of the endoscope.
10. Achalasia or any other severe esophageal motility disorder
11. Severe coagulopathy.
12. Insulin-dependent diabetes (either Type 1 or Type 2) or a significant likelihood of requiring insulin treatment in the following 12 months or a HgbA1C >= 9.
13. Subjects with any serious health condition unrelated to their weight that would increase the risk of endoscopy
14. Chronic abdominal pain
15. Motility disorders of the GI tract such as gross esophageal motility disorders, gastroparesis or intractable constipation
16. Hepatic insufficiency or cirrhosis
17. Use of an intragastric device prior to this study due to the increased thickness of the stomach wall preventing effective suturing.
18. Active psychological issues preventing participation in a life-style modification program as determined by a psychologist
19. Patients unwilling to participate in an established medically-supervised diet and behavior modification program, with routine medical follow-up.
20. Patients receiving daily prescribed treatment with high dose aspirin (> 80mg daily), anti-inflammatory agents, anticoagulants or other gastric irritants.
21. Patients who are unable or unwilling to take prescribed proton pump inhibitor medication
22. Patients who are pregnant or breast-feeding.
23. Subjects with Severe cardiopulmonary disease or other serious organic disease which might include known history of coronary artery disease, Myocardial infarction within the past 6 months, poorly-controlled hypertension, required use of NSAIDs
24. Subjects taking medications on specified hourly intervals that may be affected by changes to gastric emptying, such as anti-seizure or anti-arrhythmic medications
25. Subjects who are taking corticosteroids, immunosuppressants, and narcotics
26. Subjects who are taking diet pills
27. Symptomatic congestive heart failure, cardiac arrhythmia or unstable coronary artery disease.
28. Pre-existing respiratory disease such as chronic obstructive pulmonary disease (COPD), pneumonia or cancer.
29. Diagnosis of autoimmune connective tissue disorder (e.g. lupus, erythematous, scleroderma) or immunocompromised.
30. Specific diagnosed genetic disorder such as Prader Willi syndrome.
31. Eating disorders including night eating syndrome (NES), bulimia, binge eating disorder, or compulsive overeating
32. Known history of endocrine disorders affecting weight such as uncontrolled hypothyroidism.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 208 (Actual)
Dates: Start 2017-12-20 (Actual); Primary Completion 2020-10-29 (Actual); Study Completion 2021-10-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Barham K Abu Dayyeh, Principal Investigator — Mayo Clinic
Locations (9):
- United States (9):
  - Orlando Health, Orlando, Florida
  - University of Chicago, Chicago, Illinois
  - NorthShore University Health System, Evanston, Illinois
  - Johns Hopkins University, Baltimore, Maryland
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - Cornell University, New York, New York
  - Avera McKennan Hospital & University Health Center, Sioux Falls, South Dakota
  - University of Texas, Houston, Texas

REFERENCES:
- [Derived] Vargas EJ, Rizk M, Gomez-Villa J, Edwards PK, Jaruvongvanich V, Storm AC, Acosta A, Lake D, Fidler J, Bharucha AE, Camilleri M, Abu Dayyeh BK. Effect of endoscopic sleeve gastroplasty on gastric emptying, motility and hormones: a comparative prospective study. Gut. 2023 Jun;72(6):1073-1080. doi: 10.1136/gutjnl-2022-327816. Epub 2022 Oct 14. PMID 36241388
- [Derived] Abu Dayyeh BK, Bazerbachi F, Vargas EJ, Sharaiha RZ, Thompson CC, Thaemert BC, Teixeira AF, Chapman CG, Kumbhari V, Ujiki MB, Ahrens J, Day C; MERIT Study Group; Galvao Neto M, Zundel N, Wilson EB. Endoscopic sleeve gastroplasty for treatment of class 1 and 2 obesity (MERIT): a prospective, multicentre, randomised trial. Lancet. 2022 Aug 6;400(10350):441-451. doi: 10.1016/S0140-6736(22)01280-6. Epub 2022 Jul 28. PMID 35908555
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment Group: Overstitch ESG Procedure: Participants randomized to the treatment group will proceed to have the Overstitch Endoscopic Sleeve Gastroplasty (ESG) at the start of Year 1 and will undergo a standard moderate intensity life-style intervention during the first 12 months of participation. All patients undergoing ESG will go on a 6 weeks transitional diet. ESG patients will undergo a standard moderate intensity life-style intervention administered over 15 12 visits in the first year after ESG. ESG patients who have not achieved >25% EWL at the end of Year 1 will undergo a repeat upper endoscopy at 52 to 60 weeks to assess the durability of the plications. Patients will continue follow-up with a modified lifestyle intervention program administered over 6 visits in the second year
  Overstitch Endoscopic Suture System: Endoscopic Sleeve Gastroplasty (ESG), an endoscopic minimally-invasive weight loss procedure, utilizing a suturing device to reduce the stomach volume by 80% through the creation of sleeve. This is accomplished by a series of endoscopically placed stitches through the stomach wall.
  Lifestyle Intervention: Standard low-calorie diet plan and moderate intensity life-style intervention of 150 minutes of aerobic exercise per week for 12 months.
Period: Level 1: Lifestyle Modification vs ESG
Arm/Group | Control Group: Lifestyle Modification | Treatment Group: Overstitch ESG Procedure | Crossover Group: Lifestyle Intervention to ESG Procedure
Started | 123 | 85 | 0
Completed | 75 | 62 | 0
Not Completed | 48 | 23 | 0
Period: Level 2: Crossover Lifestyle to ESG
Arm/Group | Control Group: Lifestyle Modification | Treatment Group: Overstitch ESG Procedure | Crossover Group: Lifestyle Intervention to ESG Procedure
Started | 0 | 0 | 73
Completed | 0 | 0 | 72
Not Completed | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control Group: Lifestyle Modification | Treatment Group: Overstitch ESG Procedure | Crossover Group: Lifestyle Intervention to ESG Procedure | Total
Number analyzed (Participants) | 123 | 85 | 73 | 281
Age, Continuous [Median (Inter-Quartile Range); unit: years] — Population: Data collected from each study are being reported separately to avoid multi-counted participants.
  years
    Level 1: Lifestyle Modification vs ESG: number analyzed (Participants) | 123 | 85 | 0 | 208
    Level 1: Lifestyle Modification vs ESG | 46.0 [38.0 to 52.0] | 49.0 [42.0 to 56.0] |  | 46.5 [39.0 to 54.0]
    Level 2: Crossover Lifestyle to ESG: number analyzed (Participants) | 0 | 0 | 73 | 73
    Level 2: Crossover Lifestyle to ESG |  |  | 46 [40.0 to 51.0] | 46 [40.0 to 51.0]
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Data collected from each study are being reported separately to avoid multi-counted participants.
  Participants
    Level 1: Lifestyle Modification vs ESG: number analyzed (Participants) | 123 | 85 | 0 | 208
    Level 1: Lifestyle Modification vs ESG: Female | 104 | 74 |  | 178
    Level 1: Lifestyle Modification vs ESG: Male | 19 | 11 |  | 30
    Level 2: Crossover Lifestyle to ESG: number analyzed (Participants) | 0 | 0 | 73 | 73
    Level 2: Crossover Lifestyle to ESG: Female |  |  | 66 | 66
    Level 2: Crossover Lifestyle to ESG: Male |  |  | 7 | 7
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Population: Data collected from each study are being reported separately to avoid multi-counted participants.
  Participants
    Level 1: Lifestyle Modification vs ESG: number analyzed (Participants) | 123 | 85 | 0 | 208
    Level 1: Lifestyle Modification vs ESG: White | 67 | 58 |  | 125
    Level 1: Lifestyle Modification vs ESG: African American | 19 | 12 |  | 31
    Level 1: Lifestyle Modification vs ESG: Asian | 3 | 0 |  | 3
    Level 1: Lifestyle Modification vs ESG: Hispanic/Latino | 19 | 13 |  | 32
    Level 1: Lifestyle Modification vs ESG: Other | 10 | 1 |  | 11
    Level 1: Lifestyle Modification vs ESG: Deferred | 5 | 1 |  | 6
    Level 2: Crossover Lifestyle to ESG: number analyzed (Participants) | 0 | 0 | 73 | 73
    Level 2: Crossover Lifestyle to ESG: White |  |  | 40 | 40
    Level 2: Crossover Lifestyle to ESG: African American |  |  | 11 | 11
    Level 2: Crossover Lifestyle to ESG: Asian |  |  | 2 | 2
    Level 2: Crossover Lifestyle to ESG: Hispanic/Latino |  |  | 10 | 10
    Level 2: Crossover Lifestyle to ESG: Other |  |  | 6 | 6
    Level 2: Crossover Lifestyle to ESG: Deferred |  |  | 4 | 4
Region of Enrollment [Number; unit: participants] — Level 1: Lifestyle Modification vs ESG Population: Data collected from each year are being reported separately to avoid multi-counted participants.
  participants
    United States: number analyzed (Participants) | 123 | 85 | 0 | 208
    United States | 123 | 85 |  | 208
Region of Enrollment [Number; unit: participants] — Level 2: Crossover Lifestyle to ESG Population: Data collected from each year are being reported separately to avoid multi-counted participants.
  participants
    United States: number analyzed (Participants) | 0 | 0 | 73 | 73
    United States |  |  | 73 | 73

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Excess Weight Loss (EWL)
Description: Percentage of excess weight loss in participants at 12 months from randomization. Calculated as (weight loss/baseline excess weight) x 100, where weight loss is defined as follow-up weight minus the initial weight, and baseline excess weight is defined as index weight minus ideal weight X (X=25 kg/m²)
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: percentage of EWL
Arm/Group | Control Group: Lifestyle Modification | Treatment Group: Overstitch ESG Procedure | Crossover Group: Lifestyle Intervention to ESG Procedure
Number analyzed (Participants) | 110 | 77 | 72
percentage of EWL | 3.2 (18.6) | 49.2 (32.0) | 44.1 (35.7)

2. Secondary Outcome: Number of Participants With ≥25% EWL
Description: Total number of participants with ≥25% excess weight loss at 12 months from randomization
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Control Group: Lifestyle Modification | Treatment Group: Overstitch ESG Procedure | Crossover Group: Lifestyle Intervention to ESG Procedure
Number analyzed (Participants) | 110 | 77 | 72
Participants | 13 | 59 | 51

3. Secondary Outcome: Number of Participants Off Or With Reduction in Antihypertensive Medications
Description: Total number participants off or with reduction in antihypertensive medications
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Control Group: Lifestyle Modification | Treatment Group: Overstitch ESG Procedure | Crossover Group: Lifestyle Intervention to ESG Procedure
Number analyzed (Participants) | 48 | 36 | 29
Participants | 9 | 13 | 14

4. Secondary Outcome: Change in Blood Pressure
Description: Change in blood pressure measured in units of millimeters of mercury (mmHg)
Time Frame: Baseline, 12 months
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Control Group: Lifestyle Modification | Treatment Group: Overstitch ESG Procedure | Crossover Group: Lifestyle Intervention to ESG Procedure
Number analyzed (Participants) | 72 | 58 | 50
mmHg
  Systolic | -0.7 (14.5) | -5.2 (16.1) | -3.5 (18.5)
  Diastolic | 0.1 (10.3) | -3.3 (12.0) | -3.0 (11.6)

5. Secondary Outcome: Change in Blood Pressure for ESG Intervention From Baseline to 24 Months
Description: Change in blood pressure for participants that received ESG intervention measured in units of millimeters of mercury (mmHg)
Time Frame: Baseline, 24 months
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Treatment Group: Overstitch ESG Procedure
Number analyzed (Participants) | 58
mmHg
  Systolic | -4.0 (16.0)
  Diastolic | -2.4 (10.0)

6. Secondary Outcome: Number of Participants Off or With Reduction in Diabetes Medications
Description: Total number of participants off or with reduction in diabetes medications
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Control Group: Lifestyle Modification | Treatment Group: Overstitch ESG Procedure | Crossover Group: Lifestyle Intervention to ESG Procedure
Number analyzed (Participants) | 27 | 13 | 14
Participants | 3 | 11 | 10

7. Secondary Outcome: Change in HgbA1c
Description: Change in HgbA1c levels
Time Frame: Baseline, 12 months
Measure: Mean (Standard Deviation); unit: Percent of Glycosylated Hemoglobin
Arm/Group | Control Group: Lifestyle Modification | Treatment Group: Overstitch ESG Procedure | Crossover Group: Lifestyle Intervention to ESG Procedure
Number analyzed (Participants) | 80 | 55 | 47
Percent of Glycosylated Hemoglobin | 0.13 (0.46) | -0.36 (0.67) | -0.4 (0.56)

8. Secondary Outcome: Change in HgbA1c for ESG Intervention From Baseline to 24 Months
Description: Change in HgbA1c levels for participants that received the ESG intervention
Time Frame: Baseline, 24 months
Measure: Mean (Standard Deviation); unit: Percent of Glycosylated Hemoglobin
Arm/Group | Treatment Group: Overstitch ESG Procedure
Number analyzed (Participants) | 45
Percent of Glycosylated Hemoglobin | -0.1 (1.0)

9. Secondary Outcome: Percentage of Total Body Weight Loss (TBWL)
Description: Percentage of total body weight loss in participants
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: percentage of TBWL
Arm/Group | Control Group: Lifestyle Modification | Treatment Group: Overstitch ESG Procedure | Crossover Group: Lifestyle Intervention to ESG Procedure
Number analyzed (Participants) | 110 | 77 | 72
percentage of TBWL | 0.8 (5.0) | 13.6 (8.0) | 12.3 (8.3)

10. Secondary Outcome: Number of Participants to Achieve ≥5% TBWL
Description: Total number of participants to achieve ≥5% total body weight loss
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Control Group: Lifestyle Modification | Treatment Group: Overstitch ESG Procedure | Crossover Group: Lifestyle Intervention to ESG Procedure
Number analyzed (Participants) | 110 | 77 | 72
Participants | 18 | 70 | 61

11. Secondary Outcome: Number of Participants to Achieve ≥10% TBWL
Description: Total number of participants to achieve ≥10% total body weight loss
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Control Group: Lifestyle Modification | Treatment Group: Overstitch ESG Procedure | Crossover Group: Lifestyle Intervention to ESG Procedure
Number analyzed (Participants) | 110 | 77 | 72
Participants | 6 | 48 | 40

12. Secondary Outcome: Esophagitis at Repeat Endoscopy
Description: Total number of participants to have esophagitis at repeat endoscopy
Time Frame: 12 months
Population: Those ESG patients who have achieved >25% EWL at the end of Level 1 will not undergo a repeat endoscopy and will continue to follow-up with a lifestyle intervention in Level 2. Those ESG patients who have not achieved >25% EWL at the end of Level 1 will undergo a repeat upper endoscopy at 52
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Group: Overstitch ESG Procedure
Number analyzed (Participants) | 18
Participants | 0

13. Secondary Outcome: Change in Impact of Weight on Quality of Life-Lite (IWQOL-Lite)
Description: Changes in impact of weight on quality of life score assessed using self-reported IWQOL-lite questionnaire consisting of five domains: physical function (11 items, score range from 11-55 with higher scores indicating more negative outcome), self-esteem (7 items, score range from 7-35 with higher scores indicating more negative outcome), sexual life (4 items, score range from 4-20 with higher scores indicating more negative outcome), public distress (5 items, score range from 5-25 with higher scores indicating more negative outcome), and work (4 items, score range from 4-20 with higher scores indicating more negative outcome).
Time Frame: Baseline, 12 months
Population: Not all participants provided answers to all the domains of the Impact of Weight on Quality of Life-Lite (IWQOL-Lite) questionnaire
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control Group: Lifestyle Modification | Treatment Group: Overstitch ESG Procedure | Crossover Group: Lifestyle Intervention to ESG Procedure
Number analyzed (Participants) | 86 | 65 | 58
score on a scale
  Physical Function (11 items) | -2.5 (6.6) | -12.0 (7.4) | -8.6 (6.9)
  Self-Esteem (7 items): number analyzed (Participants) | 86 | 64 | 58
  Self-Esteem (7 items) | -1.6 (5.2) | -9.2 (7.1) | -7.8 (6.7)
  Sexual Life (4 items): number analyzed (Participants) | 84 | 63 | 57
  Sexual Life (4 items) | -1.4 (3.9) | -4.2 (4.1) | -2.6 (3.5)
  Public Distress (5 items): number analyzed (Participants) | 86 | 64 | 57
  Public Distress (5 items) | -0.9 (3.2) | -2.5 (2.9) | -1.8 (3.1)
  Work Results (4 items): number analyzed (Participants) | 86 | 64 | 57
  Work Results (4 items) | -0.3 (2.7) | -2.2 (2.7) | -1.9 (2.8)

14. Secondary Outcome: Changes in Health Status Survey Scores
Description: Changes in subject's view of health assessed using self-reported SF-36 Health Status Survey consisting of 8 scaled scores: physical function (10-items, score range from 0-100 with higher scores indicating more positive outcome), role limitations due to physical health (4-items, score range from 0-100 with higher scores indicating more positive outcome), role limitations due to emotional problems (3-item, score range from 0-100 with higher scores indicating more positive outcome), energy/fatigue (4-items, score range from 0-100 with higher scores indicating more positive outcome), emotional well-being (5-items, score range from 0-100 with higher scores indicating more positive outcome), social functioning (2-items, score range from 0-100 with higher scores indicating more positive outcome), pain (2-items, score range from 0-100 with higher scores indicating more positive outcome), general health (5-items, score range from 0-100 with higher scores indicating more positive outcome)
Time Frame: Baseline, 12 months
Population: Not all participants provided answers to all the domains of the SF-36 Health Status Survey questionnaire
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control Group: Lifestyle Modification | Treatment Group: Overstitch ESG Procedure | Crossover Group: Lifestyle Intervention to ESG Procedure
Number analyzed (Participants) | 86 | 65 | 58
score on a scale
  Physical Functioning: number analyzed (Participants) | 86 | 64 | 58
  Physical Functioning | 2.1 (25.5) | 18.9 (26.9) | 18.4 (22.5)
  Physical Health: number analyzed (Participants) | 86 | 64 | 58
  Physical Health | 4.9 (37.7) | 18.4 (33.7) | 15.1 (31.0)
  Emotional Problems: number analyzed (Participants) | 86 | 64 | 58
  Emotional Problems | -0.8 (30.7) | 4.7 (30.8) | 8.6 (30.3)
  Energy/Fatigue | 9.0 (18.5) | 14.1 (26.1) | 13.0 (20.0)
  Emotional Well-Being | 2.1 (13.2) | 1.5 (18.5) | 4.6 (14.5)
  Social Functioning: number analyzed (Participants) | 86 | 64 | 57
  Social Functioning | 3.2 (18.3) | 9.0 (29.2) | 8.8 (20.0)
  Pain | 4.4 (21.5) | 10.1 (17.6) | 7.3 (23.0)
  General Health: number analyzed (Participants) | 86 | 62 | 58
  General Health | 4.0 (14.7) | 20.4 (19.2) | 12.6 (14.5)

15. Secondary Outcome: Number of Participants With Major Depression or Severe Major Depression at Baseline
Description: Number of participants to identify with major or severe major depression measured using the self-reported Patient Health Questionnaire (PHQ-9). The PHQ-9 is self-reported 9-item questionnaire to assess degree of depression severity with total score range from 0-27 categories were defined as followed: minimal, score < 10; major depression, 10 ≤ score < 20; severe major depression, x ≥ 20
Time Frame: Baseline
Measure: Count of Participants; unit: Participants
Arm/Group | Control Group: Lifestyle Modification | Treatment Group: Overstitch ESG Procedure | Crossover Group: Lifestyle Intervention to ESG Procedure
Number analyzed (Participants) | 108 | 75 | 71
Participants
  Number with Major Depression | 14 | 7 | 9
  Number with Severe Major Depression | 2 | 1 | 1

16. Secondary Outcome: Number of Participants With Major Depression or Severe Major Depression at 12 Months
Description: as for outcome 15
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Control Group: Lifestyle Modification | Treatment Group: Overstitch ESG Procedure | Crossover Group: Lifestyle Intervention to ESG Procedure
Number analyzed (Participants) | 88 | 67 | 59
Participants
  Number with Major Depression | 10 | 2 | 1
  Number with Severe Major Depression | 2 | 0 | 0

17. Secondary Outcome: Change in Eating Behaviors
Description: Change in eating behaviors evaluated using the self-reported Three Factor Eating Questionnaire (TFEQ) consisting of 3 domains: cognitive restraint (6-items, score range from 0-100 with higher score indicating more restraint), uncontrolled eating (9-items, score range from 0-100 with lower score indicating more control), and emotional eating (3-items, score range 0-100 with higher score indicating eating with negative emotions)
Time Frame: Baseline, 12 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control Group: Lifestyle Modification | Treatment Group: Overstitch ESG Procedure | Crossover Group: Lifestyle Intervention to ESG Procedure
Number analyzed (Participants) | 86 | 64 | 58
score on a scale
  Cognitive Restraint | 4.6 (17.6) | 12.6 (19.5) | 6.0 (18.1)
  Uncontrolled Eating | -8.7 (18.0) | -14.4 (23.4) | -10.4 (16.1)
  Emotional Eating | -6.7 (23.5) | -18.3 (29.8) | -7.7 (24.0)

ADVERSE EVENTS:
Time Frame: Adverse events were collected from baseline to end of study participation for a total of approximately 2 years on all participants
Arm/Group | Control Group: Lifestyle Modification | Treatment Group: Overstitch ESG Procedure | Crossover Group: Lifestyle Intervention to ESG Procedure
All-Cause Mortality (participants affected / at risk) | 0/110 | 0/77 | 0/73
Serious Adverse Events (participants affected / at risk) | 1/110 | 12/77 | 4/73
Other Adverse Events (participants affected / at risk) | 46/110 | 77/77 | 64/73
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Control Group: Lifestyle Modification (N=110) | Treatment Group: Overstitch ESG Procedure (N=77) | Crossover Group: Lifestyle Intervention to ESG Procedure (N=73)
Abdominal Pain (Gastrointestinal disorders) | 1 (1) | 3 (3) | 0 (0)
Abscess intra abdominal (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Bloody Stool (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Bowel impaction (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Broken Hip (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Chest Pain (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
ED Visit-Sore Throat (General disorders) | 0 (0) | 1 (1) | 0 (0)
ER Visit-Coffee ground emesis (General disorders) | 0 (0) | 1 (1) | 0 (0)
ER Visit-Dehydration (General disorders) | 0 (0) | 1 (1) | 0 (0)
Esophageal mucosal tear due to device malfunction (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Gangrenous cholecystitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Headache/migraine (General disorders) | 0 (0) | 1 (1) | 0 (0)
Hospitalization-Cellulitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Hospitalization-Mental Health (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Hospitalization-Obstruction Intestinal (HCC) (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Malnutrition (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Motor Vehicle Accident (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Nausea (General disorders) | 0 (0) | 2 (2) | 0 (0)
Nausea and vomiting (General disorders) | 0 (0) | 1 (1) | 0 (0)
Pleural effusion (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Post ESG Hospital Stay (General disorders) | 0 (0) | 0 (0) | 1 (1) — Hospital stay past allotted 23 hours due to nausea
Readminission (General disorders) | 0 (0) | 0 (0) | 1 (1) — Readmission post procedure due to nausea/vomiting
Vomiting (General disorders) | 0 (0) | 2 (2) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Control Group: Lifestyle Modification (N=110) | Treatment Group: Overstitch ESG Procedure (N=77) | Crossover Group: Lifestyle Intervention to ESG Procedure (N=73)
Abdominal Pain (Gastrointestinal disorders) | 7 (8) | 56 (87) | 46 (60)
Abdominal Pain/Epigastric Pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Abdominal Spasm (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Allergic Reaction (Immune system disorders) | 1 (1) | 3 (3) | 0 (0)
Anemia (Metabolism and nutrition disorders) | 2 (2) | 2 (2) | 1 (1)
Apnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Back and Pelvic Spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Back Pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 2 (3) | 1 (1)
Bilateral Calf Discomfort (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Bilateral Frozen Shoulder (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Biliary Dyskinesia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Bladder Spasms (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Bloating (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0)
Bloody Stool (Gastrointestinal disorders) | 1 (1) | 7 (9) | 0 (0)
Blurred Vision (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1)
Burning (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Burping (General disorders) | 1 (1) | 1 (1) | 1 (1)
Calculus of Gallbladder (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Chest Pain (Cardiac disorders) | 1 (1) | 3 (3) | 0 (0)
Chest Tightness (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Chills (General disorders) | 0 (0) | 1 (1) | 0 (0)
Clinically abnormal lab findings (General disorders) | 4 (10) | 15 (36) | 5 (6)
Cold Sore (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Common Cold (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2) | 0 (0)
Concentrated Urine (Renal and urinary disorders) | 2 (2) | 19 (25) | 4 (5)
Constipation (Gastrointestinal disorders) | 10 (13) | 48 (92) | 31 (40)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1) | 2 (2)
Cough, Sore Throat, Congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
COVID-19 (Infections and infestations) | 1 (1) | 7 (7) | 1 (1)
Dark Stools (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Dehydration (Gastrointestinal disorders) | 0 (0) | 5 (7) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 10 (13) | 22 (33) | 13 (15)
Diarrhea, Nausea, Chills, Weakness, Muscle Aches (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 3 (3) | 28 (36) | 19 (22)
Ear Infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Ear Pain (Ear and labyrinth disorders) | 0 (0) | 2 (2) | 0 (0)
Edema (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Epigastric Pain (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0)
Eructation (Gastrointestinal disorders) | 4 (4) | 49 (77) | 29 (36)
Eye Hemorrhage (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Eye Laceration (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Fatigue/Lethargy (General disorders) | 2 (2) | 4 (4) | 0 (0)
Fever (Infections and infestations) | 3 (4) | 3 (3) | 0 (0)
Fibromyalgia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Finger Injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Finger Laceration (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Flu (Infections and infestations) | 2 (2) | 0 (0) | 2 (2)
Foot Infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Foot Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 1 (1)
Foot Sprain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Frozen Shoulder (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Gagging on Uvula (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Gas Pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 2 (2)
Gel tear in eye (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Groin Pull (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Hair Loss (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Halitosis (Gastrointestinal disorders) | 3 (3) | 20 (23) | 13 (13)
Hand and Leg Tremors (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Headache/Migraine (Nervous system disorders) | 14 (19) | 36 (65) | 19 (26)
Heartburn (Gastrointestinal disorders) | 17 (22) | 44 (78) | 21 (28)
Heartburn/Reflux (Gastrointestinal disorders) | 0 (0) | 2 (3) | 0 (0)
Heart Murmer (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Hiccups (Gastrointestinal disorders) | 1 (1) | 22 (33) | 13 (14)
Insomnia (Psychiatric disorders) | 2 (2) | 0 (0) | 0 (0)
Intraoperative Bleeding (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Irregular Menstrual Bleeding (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Joint and Muscle Tenderness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Joint Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Knee Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) | 1 (1)
Knee Replacement (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1)
Left Lower Quadrant Abdominal Pain (Gastrointestinal disorders) | 0 (0) | 4 (4) | 0 (0)
Left Upper Quadrant Pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Loss of Taste/Smell (General disorders) | 0 (0) | 1 (1) | 1 (1)
Lower Extremity Redness (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) — possibly due to bug bite
Lumpectomy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Lyme Disease (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Lymphedema (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Mediastinal Lymphadenopathy (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Memory Loss (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Metallic Taste in Mouth (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Motor Vehicle Accident (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Muscle Aches (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 7 (7) | 56 (90) | 42 (48)
Nausea & Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Nausea and Stomach Ache (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Nausea and Vomiting (Gastrointestinal disorders) | 0 (0) | 4 (4) | 1 (1)
Neck Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Night Sweats (General disorders) | 0 (0) | 1 (1) | 0 (0)
Oral Thrush (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Palpitations (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Parotid Salivary Gland Obstruction (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1)
Pelvic Pain (Reproductive system and breast disorders) | 3 (3) | 0 (0) | 0 (0)
Pinched Nerve in Neck (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
Pus in Old Wound Site (abdominal) (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 2 (2)
Rectal Bleeding (Gastrointestinal disorders) | 0 (0) | 3 (3) | 0 (0)
Recurrent Abdominal Abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
RLQ Abdominal Pain (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Right Finger Redness (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) — Possible bug bite
Runny Nose (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
RUQ Pain (Gastrointestinal disorders) | 0 (0) | 2 (4) | 1 (1)
Shakiness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Shin Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Shortness of Breath (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 4 (4) | 0 (0)
Shoulder Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 4 (5) | 0 (0)
Sore Throat (Infections and infestations) | 3 (3) | 1 (1) | 2 (2)
Sprained Ankle (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Stiffness, Bruising, Soreness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Strep Throat (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Syncope (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 2 (2) | 0 (0)
Tailor's Bunion of Right Foot (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Tingling Down Arms and Shoulders (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Tinnitis (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1)
Toe Fungus (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Tonsillitis (General disorders) | 0 (0) | 0 (0) | 1 (1)
Tremor (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
Umbilical Discomfort (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Upper Respiratory Infection (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0)
Urinary Retention (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
UTI (Renal and urinary disorders) | 1 (1) | 2 (3) | 2 (2)
Urine Frequency/Urgency (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Virus (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Vaginal Bleeding (2nd time) (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 40 (56) | 30 (35)
Weakness (General disorders) | 1 (1) | 0 (0) | 0 (0)
White Tongue (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Xyphoid Process Pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-11-05): https://cdn.clinicaltrials.gov/large-docs/75/NCT03406975/Prot_SAP_000.pdf